CLINICAL TRIAL: NCT04969068
Title: The Median Effective Dose of Remimazolam for Duodenoscopy Insertion During ERCP With Alfentanil 10µg/kg
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Director, Tianjin Nankai Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TianjinNK RM007
Record Dates: First submitted 2021-07-04; First posted 2021-07-20 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Anesthesia
Keywords: remimazolam; alfentanil; duodenoscopy insertion; ERCP
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The median effective dose of remimazolam for duodenoscopy insertion with alfentanil 10µg/kg (Experimental): The first patient was tested at 0.2mg/kg remimazolam (0.025mg/kg as a step size).The response of the patients to the duodenoscopy insertion during ERCP was categorized as either 'success (no movement)' or 'failure (movement)'
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Interventions:The dose of remimazolam for each patient was determined by the response of the previously tested patients using the modified Dixon's up-and-down method.The first patient was tested at 0.2mg/kg remimazolam (0.025mg/kg as a step size). Duodenoscopy insertion was conducted when MOAA/S≤1.The response of the patients to the duodenoscopy insertion during ERCP was categorized as either 'success (no movement)' or 'failure (movement).' Movement was defined as duodenoscopy insertion a failure was as gross purposeful muscular movement, coughing or vomiting occurring during or within 2 minutes of insertion of duodenoscopy. No movement was depicted when the reactions mentioned earlier were absent. If BIS>75 and MOAA/S > 1 when 3 min after the intravenous injection of remimazolam, it was considered a failure, and the patient received rescue sedation.

SUMMARY:
Remimazolam has shown promising results for sedation in colonoscopy . Alfentanil is widely used in the analgesia of ERCP . The purpose of the study was to determine the median effective dose of remimazolam for duodenoscopy insertion during ERCP with alfentanil 10µg/kg.

DETAILED DESCRIPTION:
1. Title:The median effective dose of remimazolam for duodenoscopy insertion during ERCP with alfentanil 10µg/kg.
2. Research center: Single center.
3. The population of the study: Age is between 18 and 85 years; ASA I andIII levels; Patients undergone elective ERCP surgery, non-intubation patients;
4. Sample size:The sample size was decided based on that of prior literature, which had demonstrated that at least six independent pairs with success/failure duodenoscopy insertion during ERCP are required for reliable estimates of the ED50 of remimazolam with the Dixon's up-and-down method, and data from seven independent pairs of patients were collected for this study. The ED50 (95% confidence interval, CI) of remimazolam for successful duodenoscopy insertion during ERCP was calculated according to the formula of Dixon and Massey.

6. Interventions:The dose of remimazolam for each patient was determined by the response of the previously tested patients using the modified Dixon's up-and-down method.The first patient was tested at 0.2mg/kg remimazolam (0.025mg/kg as a step size). Duodenoscopy insertion was conducted when MOAA/S≤1.The response of the patients to the duodenoscopy insertion during ERCP was categorized as either 'success (no movement)' or 'failure (movement).' Movement was defined duodenoscopy insertion a failure was as gross purposeful muscular movement, coughing or vomiting occurring during or within 2 minutes of insertion of duodenoscopy. No movement was depicted when the reactions mentioned earlier were absent.If BIS>75 and MOAA/S > 1 when 3 min after the intravenous injection of remimazolam, it was considered a failure, and the patient received rescue sedation..

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 85 years
* ASA I and III, levels;
* Patients undergone elective ERCP surgery, non-intubation patients;

Exclusion Criteria:

* Chronic pain with long-term use of analgesics, psychotropic substances (including opioids, NSAIDs, sedatives, antidepressants), alcohol abusers, with known drug allergy;
* BMI<18,BMI>30
* Abnormal renal function (BUN or Cr ) ;
* Previous abnormal surgical anesthesia recovery history;
* Hypertension or systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 95 mmHg when the patient admission to the operating room
* Suffering from esophageal reflux; • Sedatives, analgesics and antipruritic drugs were used 24 hours before operation;
* Expected difficult intubation ;
* Liver surgery history;
* Opioids allergy history;
* Take monoamine oxidase inhibitor or antidepressant within 15 days;
* COPD;
* Pregnant or parturient women;
* Involved in other drug trials within three months;
* Patients who can not communicate well with the researcher

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-23 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of success duodenoscopy insertion | 1 day
  success duodenoscopy insertion is defined by no body movement

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Nankai Hospital, Tianjin, Tianjin Municipality, China